CLINICAL TRIAL: NCT07280351
Title: Duraplasty for Acute Traumatic Spinal Cord Injury
Acronym: DATSCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-42716; CDMRP-SC240090 (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injury, Acute; Spinal Cord Injury (SCI), Initial Encounter; Spinal Cord Injury Cervical
Keywords: spinal cord injury; SCI; expansile duraplasty; duraplasty; acute SCI; traumatic SCI; acute traumatic spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental (Experimental): Participants in this arm receive expansile duraplasty during their standard surgery for spinal cord injury.
  Interventions: Procedure: Expansile duraplasty
- Control (No Intervention): Participants in this arm do not receive expansile duraplasty during their standard surgery for spinal cord injury.

INTERVENTIONS:
Procedure: Expansile duraplasty — During their standard of care surgery, in participants undergoing expansile duraplasty, the dura of the spinal cord will be opened linearly at midline to a target length of 3.5cm during surgery and a 1.5 wide x 3.5cm long suturable dural patch will be sutured in place with 6-0 polypropylene running suture to expand the intrathecal space and create room for post-injury spinal cord swelling. Duraplasty is performed during the index surgery for traumatic spinal cord injury, not as a separate, nor delayed surgery. The pia and the spinal cord will not be opened.
  Arms: Experimental

SUMMARY:
The goal of this clinical trial is to learn if a procedure called "expansile duraplasty" can improve recovery in adults who have experienced an acute traumatic spinal cord injury (SCI). The main questions it aims to answer are:

* Does expansile duraplasty work to improve recovery in people with acute traumatic SCI?
* How safe is the use of expansile duraplasty in people with acute traumatic SCI?

Researchers will compare the strength, movement, and overall recovery of participants who receive expansile duraplasty to that of participants who do not receive expansile duraplasty to see if the use of expansile duraplasty leads to better recovery for people with acute traumatic SCI.

Participants will be randomly placed in one of two groups: an Experimental group and a Control group. Participants in the Experimental group will receive expansile duraplasty during their standard SCI surgery. Participants in the Control group will not receive expansile duraplasty during their standard SCI surgery. All participants will:

* Provide samples of blood and cerebrospinal fluid
* Undergo magnetic resonance imaging (MRI) scans
* Undergo an assessment of the ability to move arms/legs and feel touch or pin prick
* Answer questionnaires about medical history, pain, health, and independence with activities of daily living

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, single-blinded controlled trial aimed at evaluating safety and effectiveness of expansile duraplasty in people hospitalized for acute traumatic spinal cord injury (SCI).

Traumatic SCI remains a challenging clinical problem for which treatment options remain limited, despite significant ongoing efforts by industry, non-profit organizations and academia to unveil the mechanisms behind it. There is currently no clearly beneficial pharmaceutical therapy for SCI, so in the absence of suitable pharmacotherapy, early surgical decompression and optimization of spinal cord perfusion have been emerged as targets for intervention. Common surgical techniques do not address intrathecal compression due to spinal cord swelling. The lack of dural decompression after SCI is in contrast to traumatic brain injury, where dural opening is a routine part of decompressive craniectomy. There remains a paucity of data on whether durotomy or expansile duraplasty may provide additional benefit in decompressing the injured spinal cord, though preclinical animal data has for decades been in favor of early decompression, and there is evidence from non-randomized human studies that suggest duraplasty may lead to improved outcomes for SCI patients. These data, along with other published SCI research, served as motivation to explore expansile duraplasty in humans.

Specific objectives of this randomized clinical trial are to evaluate (i) effectiveness of the expansile duraplasty in improving neurologic motor outcomes in patients with acute traumatic SCI; (ii) safety of expansile duraplasty in acute traumatic SCI patients; (iii) exploratory effectiveness of reducing intrathecal pressure (ITP) by expansile duraplasty in patients with acute traumatic SCI.

Eligible patients admitted at participating sites will be approached for study participation prior to their standard of care (SOC) index surgery for acute traumatic SCI. Consenting participants will be randomized into either the Experimental or Control group, and those in the Experimental group will receive expansile duraplasty during their SOC surgery. A blood sample, cerebrospinal fluid (CSF) sample, motorsensory assessment, and magnetic resonance imaging (MRI) scan will be obtained pre-operatively. Additional CSF samples, motorsensory assessments, and MRI scan will be obtained post-operatively during participants' subsequent stay in the intensive care unit (ICU) and acute care units. During this stay, participants will receive standard of care medical treatment for SCI that is standardized across all sites (except where specified), including: close monitoring, including hemodynamic and pressure monitoring; intrathecal pressure measurement, at least once hourly for five days; maintenance of spinal cord perfusion pressure (SCPP) at 65 and above, via vasopressor administration as needed, for at least five days; post-treatment rehabilitation and occupational therapy procedures, per standard of care at the investigational site. During this time also, the participants will be monitored for Adverse Events (AEs). Questionnaires will be administered and clinical information such as injury characteristics, vitals measurements, and lab results will be collected during the participants' hospital stay.

Study follow-up visits occur at 6 and 12 months post-injury, with the primary endpoint at the 6-month follow-up. At the follow-up visits, vitals will be measured, a motorsensory assessment completed, and questionnaires on pain and quality of life will be administered. The Investigator will assess participants at each study visit for the occurrence of AEs.

ELIGIBILITY:
Inclusion Criteria:

* In initial hospitalization for recent (less than 24 hours) acute, traumatic spinal cord injury at a participating site
* Diagnosis of acute, traumatic spinal cord injury
* AIS grade A - C
* C3 - C7 neurological level of injury on ISNCSCI exam
* Imaging showing cord compression
* Surgical decompression initiated within 24 hours after injury
* At sites where lumbar drain placement is standard of care: placement of lumbar drain
* Able to cooperate in the completion of standardized neurological examinations

Exclusion Criteria:

* Injury arising from penetrating mechanism
* Pregnancy
* In custody
* Under psychiatric hold
* Presence of traumatic durotomy severe enough to preclude study treatment or procedures, in the opinion of the treating surgeon
* Extensive polytrauma as determined by ISS score of >25
* History of prior spinal cord injury
* Concomitant non-traumatic spinal cord injury (e.g. infection or tumor)
* Significant concomitant head injury as defined by a Glasgow Coma Scale (GCS) <14 or a clinically significant abnormality on a head CT (head CT required only for patients suspected to have a brain injury at the discretion of the investigator)
* GCS Motor score < 6
* Pre-existing neurologic or mental disorder which would preclude accurate evaluation and follow-up (i.e. Alzheimer's disease, Parkinson's disease, unstable psychiatric disorder with hallucinations and/or delusions or schizophrenia)
* The treating surgeon deems that an anterior-only approach to decompression and/or stabilization (e.g. anterior cervical discectomy and fusion) is the best treatment plan based on the patient's injury pattern
* Recent history (less than 1 year) of chemical substance dependency or significant psychosocial disturbance that may impact the outcome or study participation, in the opinion of the investigator
* Active malignancy or history of invasive malignancy within the last five years, with the exception of superficial basal cell carcinoma or squamous cell carcinoma of the skin that has been definitely treated. Patients with carcinoma in situ of the uterine cervix treated definitely more than 1 year prior to enrollment may enter the study.
* Thrombocytopenia, defined as less than 100,000 platelets per microliter of blood, that is not correctible by transfusion
* Coagulopathy, defined as INR > 1.4, that is not correctible by transfusion
* Allergy to the study material, which may include fetal bovine tissue and collagen.
* Contraindications for study treatment or procedures
* Unable to give informed consent prior to their standard of care surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Change in AIS grade from baseline | From admission to 6 months post-injury
  The American Spinal Injury Association (ASIA) established the ASIA Injury Scale (AIS). The AIS grade is derived from the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) exam, ASIA's standard assessment for documentation of the level and severity of a spinal cord injury. The ISNCSCI yields a grade from A to E, wherein A indicates greater severity.

SECONDARY OUTCOMES:
SCIM III scores | At 6 months post-injury
  The Spinal Cord Independence Measure (SCIM) version III is a questionnaire that captures independence in activities of daily living following spinal cord injury. The SCIM yields a score from 0 to 100, with a higher number indicating a greater degree of independence.
SF-36 scores | At 6 months post-injury
  The 36-Item Short Form Survey (SF-36) is a 36-item patient-reported questionnaire that measures health-related quality-of-life. It covers eight health domains. Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
Pain assessment (modified from Neuropathic Pain 4; International Spinal Cord Injury Pain Basic Data Set version 2.0) | At 6 months post-injury
  The study will use a pain questionnaire modified slightly from the Neuropathic Pain 4 (DN4) assessment (which captures symptoms of neuropathic pain) and the International Spinal Cord Injury Pain Basic Data Set (ISCIPBDS) version 2.0 (which characterizes pain problems). These questions will yield quantitative and qualitative data regarding pain intensity and neuropathic symptoms, including a score of pain intensity with values ranging from 0 to 10, with 0 being "No pain" and 10 being "Pain as bad as you can imagine."
Proportion of time during first 5 days after injury that SCPP was greater than 65 mmHg | From admission to 5 days post-injury
  Spinal cord perfusion pressure (SCPP) is a measure of the pressure gradient that drives blood flow through the spinal cord. It is measured in millimeters of mercury (mmHg), and it is calculated in this study as the difference between the mean arterial pressure (MAP) and the intrathecal pressure (ITP).
Maximum Spinal Cord Compression (MSCC) metric | At 3 days post-injury
  Magnetic resonance imaging (MRI) scans are used to derive a quantitative metric of the intrathecal space calculated as: ([2 x (post-op cord diameter at injury site - pre-op diameter at injury site)/(cord diameter at segment above injury + cord diameter at segment below injury)] x 100). A value is obtained from the post-operative MRI scan performed at 3 days post-injury, and the values between the Experimental and Control groups are compared.

OTHER OUTCOMES:
Incidence of adverse events | From enrollment to 6 months post-injury
  Number of observed events following the time of intervention during a participant's standard surgery. Examples of adverse events (AE) that will be carefully monitored include: hemodynamic instability, patient condition deterioration, unanticipated AE.

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Saigal, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No